CLINICAL TRIAL: NCT06217133
Title: Heart Rate Variability of Premature Newborn Subject to Two CPAP Methods
Brief Title: Heart Rate Variability of Premature Newborn
Acronym: HRV
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Federal University of Uberlandia (Other)
Collaborators: Adriano de Oliveira Andrade (Unknown)
Responsible Party: Principal Investigator, Letícia de Queiroz Martins, Letícia de Queiroz Martins, Federal University of Uberlandia
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: Federal University Uberlandia
Record Dates: First submitted 2024-01-02; First posted 2024-01-22 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Autonomic Nervous System Imbalance
Keywords: Heart rate variability; Neonatal intensive care unit; Non-invasive ventilation
MeSH Terms: interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Intervention Model Description: The researchers will compare the conventional CPAP and bubble CPAP group according to randomization.
  The participant selected for conventional CPAP will receive conventional CPAP for 24 hours, then receive bubble CPAP for 24 hours the following day. The opposite will be done for the participant drawn for CPAP bubbles.All participants will be evaluated on two different days, on one day data collection will be carried out using conventional CPAP and on the other day bubble CPAP according to randomization. The days will be consecutive and premature babies will remain on each type of CPAP for 24 hours.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): The analysis of heart rate variability will be carried out in theIn the control group (NT), data collection will be carried out in the Rooming Room in a single reference collection lasting 20 minutes, and analyzed in 4 5-minute intervals. Newborns will be full term and will be in the supine position, lying in the common crib and resting. All collections for this group will be carried out in the afternoon on a day to be agreed with the mother or responsible companion.
- CPAP Group (Active Comparator): The analysis of heart rate variability will be carried out in the in the CPAP group, conventional and in the bubble CPAP.
  Interventions: Device: CPAP

INTERVENTIONS:
Device: CPAP — Conventional CPAP will be administered according to the unit's routine on ventilators of different brands and models according to service availability. Binary prongs, from brands available in the service, will be used as an interface without touching the nasal septum with the size recommended by the manufacturer and in accordance with the protocol established in the unit.
  TThe CPAP bubbles will be administered using the CPAP NEONATAL BABYPAP® MODEL 1150 S equipment, which is an electromedical device for non-invasive ventilatory assistance for newborns that generates continuous pressure in the airways (CPAP) controlled by means of a column of water that bubbles, through a flow of heated and humidified medical gas mixture supplied by a breathing circuit to the patient's nasal passage.
  Other Names: continuous positive airway pressure
  Arms: CPAP Group

SUMMARY:
To analyze the effects of two CPAP methods on the HRV of PTNBs during their routine routine in the HCUFU neonatal ICU. This is a randomized clinical trial, with controlled groups and cross over with healthy term newborns (RNT) as a control group admitted to the HC-UFU rooming-in and premature newborns (PTRN), between 28 and 32 weeks pregnant women with nasal CPAP group admitted to the neonatal ICU of the same hospital. The HRV recorded by the POLAR® RS800cx cardiac monitor will be analyzed, with a sampling rate of 1000 Hz.

The main question[s] it aims to answer are:

* Is there a difference in heart rate variability between newborns using conventional nasal CPAP and nasal bubble CPAP?
* Is it possible to conclude that one of the methods has a greater sympathetic or parasympathetic tone compared to the other?

Premature participants will be in the incubators in a supine position with 30 minutes rest after the last handling. Each data collection will last 60 minutes and will be carried out three times a day in the morning, afternoon and night shifts, for each 1-hour collection, HRV will be analyzed in 12 5-minute intervals, establishing an average for each variable of the data. HRV during a 1-hour period.

The researchers will compare the conventional CPAP and bubble CPAP group according to randomization.

* In the control group, data collection will be carried out in the Rooming Room in a single reference collection lasting 20 minutes, and analyzed in 4 5-minute intervals.
* The participant selected for conventional CPAP will receive conventional CPAP for 24 hours, then receive bubble CPAP for 24 hours the following day. The opposite will be done for the participant drawn for CPAP bubbles.

The comparison between the conventional CPAP and bubble CPAP groups will occur to find out whether it is possible to identify the type of non-invasive ventilation that allows an increase in HRV and parasympathetic tone variables, as well as a reduction in sympathetic tone variables and the stress index of premature babies.

ELIGIBILITY:
Inclusion Criteria:

* All preterm infants between 28 and 32 weeks of gestation using nasal CPAP and who are at least 8 and at most 12 days old will be included in the study.

Exclusion Criteria:

* hemodynamic instability,
* hydroelectrolyte disorders that influence cardiac function,
* post-operative,
* congenital abnormalities,
* pulmonary hypertension,
* decompensated ductus arteriosus,
* untreated atelectasis,
* pneumothorax,
* newborns who are using drains, whether chest or abdominal,
* presence of necrotizing enterocolitis
* grade 3 nasal septum injury,
* signal captured without the necessary quality to be used in research,
* premature babies who, for whatever reason, do not have two collections carried out on consecutive days until the twelfth day of life.

Ages: 28 Weeks to 32 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 65 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
HRV variables in time domains | A total of two evaluation days will be carried out, which will be divided into: 1 full hour in the morning, afternoon and evening, totaling 3 hours for each consecutive evaluation day
  The time domain variables are:
  average of RR intervals (Mean RR) expressed in milliseconds (ms); average beats per minute (Mean HR) expressed in (bpm); standard deviation of all normal RR intervals (SDNN) expressed in (ms); square root of the mean square differences between successive RR intervals (RMSSD) expressed in (ms); percentage of adjacent RR intervals with a difference in duration greater than 50 ms (pNN50) expressed in percentage (%).
Frequency domain variables | A total of two evaluation days will be carried out, which will be divided into: 1 full hour in the morning, afternoon and evening, totaling 3 hours for each consecutive evaluation day
  The frequency domain variables are:
  very low frequency (VLF) expressed in hertz (Hz); low frequency (LF) expressed in Hz; high frequency (HF) expressed in Hz.
The non-linear parameters of heart rate variability | total of two evaluation days will be carried out, which will be divided into: 1 full hour in the morning, afternoon and evening, totaling 3 hours for each consecutive evaluation day
  The non-linear parameters of heart rate variability are:
  short-term (instantaneous) beat-to-beat RR variability of the Poincaré plot (SD1) expressed in milliseconds (ms); long-term (continuous) beat-to-beat variability of the Poincaré plot (SD2) also expressed in ms and the SD2/SD1 ratio.

CONTACTS AND LOCATIONS:
Overall Officials: Lilian Rodrigues de Abreu Macedo, 3, Study Chair — Federal University of Uberlandia